CLINICAL TRIAL: NCT00440544
Title: A Phase I Trial of the Safety and Immunogenicity of an Adjuvated TB Subunit Vaccine (Ag85B-ESAT6 + LTK63) Administered at 0 and 2 Months
Brief Title: A Phase I Trial of a LTK63 Adjuvated Tuberculosis Nasal Subunit Vaccine (Ag85B-ESAT6)
Acronym: TMUVA-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety Issues
Sponsor: St George's, University of London (Other)
Collaborators: Statens Serum Institut (Other); Novartis Vaccines (Industry); European Union (Other)
Responsible Party: David JM Lewis, Principal Investigator, SGUL
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMUVA-01; EudraCT Number: 2005-005140-81; FP6-2002-LIFESCIHEA-2.3 503240
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; vaccine; nasal immunization
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): 100 ug H1 antigen alone in BCG naive subjects
  Interventions: Biological: Ag85B-ESAT6 fusion protein H1
- 2 (Experimental): 100 ug H1 antigen + LTK63 adjuvant 30 ug in BCG naive subjects
  Interventions: Biological: Ag85B-ESAT6 fusion protein H1
- 3 (Experimental): 50 ug H1 antigen in BCG immunized subjects
  Interventions: Biological: Ag85B-ESAT6 fusion protein H1
- 4 (Experimental): 50 ug H1 antigen + LTK63 adjuvant 30 ug in BCG immunized subjects
  Interventions: Biological: Ag85B-ESAT6 fusion protein H1
- 5 (Experimental): 100 ug H1 antigen in BCG immunized subjects
  Interventions: Biological: Ag85B-ESAT6 fusion protein H1
- 6 (Experimental): 100 ug H1 antigen + LTK63 adjuvant 30 ug in BCG immunized subjects
  Interventions: Biological: Ag85B-ESAT6 fusion protein H1

INTERVENTIONS:
Biological: Ag85B-ESAT6 fusion protein H1 — 100 ug H1 antigen in BCG naive subjects
  Arms: 1
Biological: Ag85B-ESAT6 fusion protein H1 — 100 ug H1 antigen + LTK63 adjuvant 30 ug in BCG naive subjects
  Arms: 2
Biological: Ag85B-ESAT6 fusion protein H1 — 50 ug H1 antigen in BCG immunized subjects
  Arms: 3
Biological: Ag85B-ESAT6 fusion protein H1 — 50 ug H1 antigen + LTK63 adjuvant 30 ug in BCG immunized subjects
  Arms: 4
Biological: Ag85B-ESAT6 fusion protein H1 — 100 ug H1 antigen in BCG immunized subjects
  Arms: 5
Biological: Ag85B-ESAT6 fusion protein H1 — 100 ug H1 antigen + LTK63 adjuvant 30 ug in BCG immunized subjects
  Arms: 6

SUMMARY:
The purpose of this study is to determine whether a subunit tuberculosis vaccine given as two nasal immunizations composed of a hybrid protein antigen from M. tuberculosis virus mixed with a toxoid adjuvant, causes untoward adverse reactions when administered to healthy adult volunteers. Both subjects who have not received Bacillus Calmette-Guerin (BCG) and subjects who have already received BCG will be enrolled. An initial evaluation of immune responses to the vaccine will also be undertaken.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a subunit tuberculosis vaccine given as two nasal immunizations composed of a hybrid protein antigen from M. tuberculosis virus mixed with a toxoid adjuvant, causes untoward adverse reactions when administered to healthy adult volunteers. Both subjects who have not received BCG and subjects who have already received BCG will be enrolled. An initial evaluation of immune responses to the vaccine will also be undertaken using flow cytometry to enumerate antigen specific IFNg containing T cells; ELISPOT to determine IFNg secreting antigen specific T cells; serology and nasal wash antibody.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy, based on medical examination at inclusion
* Male or female subjects, aged between 18 and 55 years
* Willing and likely to be able to comply with the trial procedures
* Prepared to grant authorized persons access to their medical records

Additional inclusion criterion for BCG-non-vaccinated subjects:

* BCG-non-vaccinated (i.e., absence of a BCG-scar)
* Negative Mantoux skin test

Additional inclusion criterion for BCG-vaccinated subjects:

* BCG-vaccinated (i.e., presence of a BCG-scar)

Exclusion Criteria:

* History of TB or known exposure to TB
* Radiological findings on chest X ray compatible with previous or current infection with tuberculosis
* Positive QuantiFERON® TB-Gold test Evidence of previous, current or latent tuberculosis
* Evidence of previous, current or latent tuberculosis
* History of severe organ-system diseases
* Known hypersensitivity to any of the vaccine components
* History of allergic disorders
* Vaccinated with other vaccine within 3 months before first vaccination
* Congenital and/or acquired immune diseases
* Administration of systemic immune modulating drugs (steroids, immunosuppressive drugs or immunoglobulin) within 3 months before the first vaccination (topical steroids not included)
* Autoimmune diseases
* HIV, HBV and HCV sero-positive
* Established diagnosis of a neurological or neuromuscular disease, and specifically any history of abnormality with respect to sense of smell (olfactory nerve dysfunction), or previous or current facial nerve paralysis
* Congenital or acquired abnormalities or disorders related to nasal and nasopharyngeal cavities
* Current use of any medication taken through the nasal/inhalatory route including cocaine or other drugs
* Laboratory parameters outside of normal ranges considered clinically significant
* Pregnant according to urine pregnancy test
* Females not willing to use contraceptives or who are breastfeeding
* Intake of trial medication in other clinical trials within 6 months of the first vaccination

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile (medical examinations, adverse events and laboratory safety tests) of a nasal TB subunit vaccine with and without adjuvant given as two doses with 2 months interval. | 8 months

SECONDARY OUTCOMES:
To evaluate the cell mediated and humoral immunogenicity profile of a nasal TB subunit vaccine with and without adjuvant, given as two doses with 2 months interval. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — St George's, University of London, UK
Locations (1):
- St George's Vaccine Institute, London, England, United Kingdom

REFERENCES:
- See also: St George's Vaccine Institute Home website — http://www.vaccine.ac.uk